CLINICAL TRIAL: NCT03202420
Title: Pilot Study to Test the Feasibility, Acceptability, and Weight Change of Take Off Pounds Sensibly (TOPS) in a Safety Net Clinic
Brief Title: Study to Test the Feasibility, Acceptability, and Weight Change of Take Off Pounds Sensibly (TOPS) in a Safety Net Clinic
Acronym: TOPS at DOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080518
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — TOPS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOPS (Experimental): Participants will attend weekly TOPS meetings with standard weekly weigh ins
  Interventions: Other: TOPS

INTERVENTIONS:
Other: TOPS — Take Off Pounds Sensibly (TOPS) is a national, nonprofit, peer-led, group-based, weight loss program that offers a comprehensive program on diet and physical activity with group support for weight management.

SUMMARY:
The purpose of this pilot proposal are the following: 1) to determine the feasibility and acceptability of integrating the TOPS weight loss program into underserved populations through an urban safety net clinic and 2) to gather preliminary data of weight change to inform the design of a future randomized, controlled trial to determine the efficacy of the TOPS program in safety net clinics.

To achieve these goals, the investigators will pursue the following Specific Aims:

Specific Aim 1. Assess the feasibility and acceptability of integrating the TOPS program into an urban safety net clinic, with process measures (i.e., recruitment/refusal rates and retention/dropout rates) and focus groups.

Hypothesis 1. Integrating the TOPS program into an urban safety net clinic is feasible and acceptable to participants.

Specific Aim 2. Assess the percent of participants in the TOPS intervention arm with clinically significant weight change (i.e., weight loss of ≥5% of initial body weight) at 12, 26, and 52 weeks.

Hypothesis 2. 10%, 25%, and 33% of participants in the TOPS intervention arm will lose ≥5% of initial body weight at 12, 26, and 52 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be patients of the DOC.
* BMI: Asian patients with a BMI of ≥23 kg/m2 and patients of other racial and ethnic backgrounds will be included if have a BMI of ≥25 kg/m2. Asian patients are allowed to participate at a BMI in the normal range because they are more likely to develop diabetes (or insulin resistance or glucose intolerance at a BMI of 23 kg/m2).

Exclusion Criteria:

* Mental illness that would cause disruptions to group meetings
* Cognitive impairment that would preclude participants from understanding the program
* Type 2 diabetics on insulin or sulfonylureas without provider approval
* untreated hyper- or hypothyroidism
* current cancer diagnosis
* history of cancer (other than skin cancer)
* gastrointestinal disorders affecting food intake
* use of medications thought to effect metabolism, body weight, energy expenditure, or appetite
* women currently pregnant or lactating, planning to become pregnant, or less than 6 months post-partum
* weight loss of > 5% in past 6 months
* major psychiatric disorder
* current moderate to severe symptoms of depression
* eating disorders
* current alcohol or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 12, 24, and 52 weeks
  Weekly weight data will be collected by the DOC Designee at baseline, 12, 24, and 52 weeks.

SECONDARY OUTCOMES:
Program Attendance | 52 Weeks
  Calculate the percentage of TOPS at DOC group session attendance (sessions attended/total offered).
Retention as measured by attendance sheets | 12, 24 and 52 weeks
  Calculate the retention of participants in the TOPS at DOC program at 12, 24, and 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Nia S Mitchell, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke General Internal Medicine, Durham, North Carolina, United States